CLINICAL TRIAL: NCT02235727
Title: A Phase 1, Double-Blind, Randomised, Placebo-Controlled, Study to Evaluate the Safety and Pharmacokinetics of GBR 900 in Adult Healthy Volunteers
Brief Title: Safety and Tolerability of GBR 900 in a Single Ascending Dose Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Glenmark Pharmaceuticals Ltd. India (Industry)
Collaborators: Glenmark Pharmaceuticals S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GBR 900-101; 2013-005480-31 (EudraCT Number)
Record Dates: First submitted 2014-08-07; First posted 2014-09-10 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GBR 900 (Experimental): Test treatment GBR 900
  Interventions: Drug: GBR 900
- Placebo (Placebo Comparator): Placebo Treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GBR 900
  Arms: GBR 900
Drug: Placebo
  Arms: Placebo

SUMMARY:
A Single Dose Study of GBR 900 in Healthy Volunteers.

DETAILED DESCRIPTION:
This is a phase I study of GBR 900 in healthy volunteers. The purposes of this study are to look at safety, how well the study drug is tolerated, how much of the study drug gets into the blood stream, and how long it takes the body to get rid of it when given to humans. Information about any side effects that may occur will also be collected. Each participant will remain in the study for approximately 3.5 months. This study is for research purposes only and is not intended to treat any medical condition.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) within the range 18.5-32 kg/m2 (inclusive); weight must be ≥ 50 kg.
2. Men and women aged between 18 and 55 years (inclusive). Female subjects must be of non-child-bearing potential
3. Subjects who are otherwise healthy and free from clinically significant illness or disease as determined by medical history, vital signs, physical examinations, and other tests performed by the investigator.

Exclusion Criteria:

1. Subjects with a history of neuropathy or otherwise present with risk factors for neurological toxicity like chronic alcoholism or clinically significant neurological (e.g. dementia, cognitive decline, seizure disorders) or psychiatric disorders.
2. Subjects with a recent history of live vaccination within the past 3 month or presence of active infections within the previous month.
3. Subjects with previous exposure to antibody therapies or administration of immunoglobulins (Ig) within 6 months of randomization.
4. Subjects with a history of or presence of inflammatory disease or rheumatological diseases or joint diseases including OA or any undiagnosed pain in joints.
5. Subjects with a current and/or recent history of arthralgia or a history of fibromyalgia, migraine, neuralgia, or systemic painful conditions, or medical or arthritic conditions or any undiagnosed pain or systemic inflammatory disorders.
6. Any evidence of organ dysfunction or any clinically significant deviation from the normal in history, physical or neurological determinations or investigations or has a clinical condition or receiving therapy that, in the opinion of the Investigator, would make the subjects unsuitable for study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2014-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Drug related adverse events (AEs) or any serious AEs | 71 days
  All treatment - emergent adverse events (TEAEs), occuring during the study, in terms of nature, onset, duration, severity, relationship and outcome of adverse events and serious adverse events in adult healthy volunteers from baseline to day 71.

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) of single ascending doses of GBR 900 in adult healthy volunteers | Pre-dose and post-dose at planned multiple time points from 2 hours to 168 hours and from day 15 until day 71
Area Under Curve [(AUC (0-∞) and AUC (0-t)] of single ascending doses of GBR 900 in adult healthy volunteers | Pre-dose and post-dose at planned multiple time points from 2 hours to 168 hours and from day 15 until day 71
Half life (t1/2) of single ascending doses of GBR 900 in adult healthy volunteers | Pre-dose and post-dose at planned multiple time points from 2 hours to 168 hours and from day 15 until day 71
Immunogenicity of GBR 900 | Pre-dose and at day 29, day 43, and day 71

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, MBChB, PhD, MRCS, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit Ltd, Leeds, Yorkshire, United Kingdom